CLINICAL TRIAL: NCT05378646
Title: An Open Controlled Study of the Efficacy and Safety of Ingaron (Interferon-gamma Human Recombinant) in the Treatment of Chronic Prostatitis
Brief Title: Efficiency and Safety of the Drug Ingaron (Interferon-gamma Human Recombinant) in the Treatment of Chronic Prostatitis
Acronym: ING-HP-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SPP Pharmaclon Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ING-HP-1
Record Dates: First submitted 2022-04-20; First posted 2022-05-18 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2021-11

CONDITIONS: Chronic Prostatitis
Keywords: interferon gamma; IFN-g; Chronic prostatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Patients received Ingaron 500,000 IU subcutaneously once a day, every other day. The course of treatment is 7 injections. The first injection was given on the first day of active therapy. Subsequent injections were given every other day. The period of active therapy was 14 days.
  Interventions: Drug: Interferon gamma human recombinant (IFN-G)
- Control (No Intervention): Patients received standard treatment for chronic prostatitis. The period of active therapy was 14 days.

INTERVENTIONS:
Drug: Interferon gamma human recombinant (IFN-G) — received by microbiological synthesis; specific antiviral activity on cells is 2x10*7 Units per mg of protein
  Other Names: Ingaron; Interferon gamma human recombinant
  Arms: Experimental

SUMMARY:
The primary purposes of the study are to evaluate the effectiveness of Ingaron in the complex therapy of chronic prostatitis, to assess the safety of using Ingaron in patients with chronic prostatitis.

DETAILED DESCRIPTION:
Literature data and the results of preclinical studies of interferon-gamma, as well as the features of the immunopathogenesis of chronic prostatitis, show the expediency of studying the use of Ingaron in this pathology.

The study was conducted to compare the efficacy and safety of Ingaron in combination with standard therapy with its subcutaneous administration and standard therapy in patients with chronic prostatitis.

The study was planned to include 50 male patients aged at least 18 years with a confirmed diagnosis of chronic prostatitis.

In the course of the study, Ingaron was administered at a dose of 500,000 IU once a day, every other day. In addition to Ingaron, patients received antibiotic therapy, anti-inflammatory drugs, alpha-blockers (if necessary). Magnetic laser therapy and prostate massage were also provided.

The patients were divided into 2 groups: main and control.

ELIGIBILITY:
Inclusion Criteria:

1. Age at least 18 years old (at the time of inclusion).
2. Objectively confirmed diagnosis of chronic prostatitis at the time of inclusion in the study (more than 10 leukocytes / field of view in cytological examination of prostate secretion; more than 1x10^5 CFU in bacteriological examination of prostate secretion (regardless of the nature of the inoculated microflora)).
3. Concomitant myco-, ureaplasma, gardnerella, chlamydial, urogenital viral infection is not excluded.
4. The volume of residual urine (Q max) is not more than 70 ml.
5. The maximum urination rate, according to urofluometry, is not less than 10 ml / sec.
6. Allowed previous therapy of chronic prostatitis, not less than 30 days after the end of the last course of treatment.
7. If there is a history of surgical treatment for benign prostatic hyperplasia, the time from the moment of surgery to inclusion in the study is at least 6 months.
8. Availability of written informed consent to participate in the clinical study.

Exclusion Criteria:

1. Positive test results for syphilis (Wasserman reaction), hepatitis (HbsAg, anti-HCV), HIV infection.
2. Known allergic reactions to interferons, or other significant allergic diseases.
3. A history of autoimmune disease.
4. The presence of external drains of the organs of the genitourinary system.
5. The presence of histologically proven prostate cancer.
6. A history of diabetes mellitus.
7. Any immunotropic therapy within the last 6 weeks prior to enrollment in the study.
8. Condition after organ transplantation, constant intake of immunosuppressive drugs.
9. Severe pathology from the cardiovascular system (uncontrolled arterial hypertension, unstable angina pectoris, congestive heart failure, cardiac arrhythmias), a history of myocardial infarction or cerebrovascular accident within the last 6 months.
10. Severe pathology of the liver (increased content of AST, ALT 2 times higher than the upper limit of the norm, the content of total bilirubin> 2 mg / dl), kidney (creatinine content> 1.5 mg / dl); signs of hepatic and / or renal failure.
11. Other serious (acute or chronic) pathological conditions, including mental illness, as well as abnormalities in laboratory parameters, which, in the opinion of the investigator, may increase the risk associated with participation in the study or affect the interpretation of the efficacy and safety data obtained in this research.
12. Alcohol and / or drug dependence.
13. Participation in other clinical trials in the last 3 months prior to inclusion.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-01-29 (Actual); Primary Completion 2009-12-31 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Dynamics of the total score and improvement in the quality of life on the scale IPSS. | Day 13
  The sum of points was assessed, as well as the symptom complex on the basis of the "IPSS" questionnaire - the international system for the total assessment of symptoms of prostate diseases in points (WHO, 1992). The severity of symptoms was assessed from 0 to 6 points.
  symptoms of prostate diseases in points (WHO, 1992). The severity of symptoms is rated from 0 to 6 points.
Immunohistochemical study of prostate secretion with assessment of cytological parameters. | Day 14
  Content of polymorphonuclear leukocytes in prostate secretion.
Immunohistochemical study of prostate secretion with assessment of cytological parameters. | Day 14
  The content of lymphocytes in prostate secretion.
Evaluation of cytological parameters of prostate secretion. | Day 14
  The number of lecithin grains.
Evaluation of cytological parameters of prostate secretion. | Day 14
  The number of epithelial cells.
Microscopy of prostate secretion and immunohistochemical study of prostate secretion with assessment of cytological parameters. | Day 14
  The effect of interferon-gamma on T-lymphocytes.
Evaluation of cytological parameters of prostate secretion. | Day 90
  The content of polymorphonuclear leukocytes in prostate secretion.
Immunohistochemical study of prostate secretion with assessment of cytological parameters. | Day 90
  The content of lymphocytes in prostate secretion.
Evaluation of cytological parameters of prostate secretion. | Day 90
  The number of lecithin grains.
Evaluation of cytological parameters of prostate secretion. | Day 90
  The number of epithelial cells.
Microscopy of prostate secretion and immunohistochemical study of prostate secretion with assessment of cytological parameters. | Day 90
  The effect of interferon-gamma on T-lymphocytes.
Evaluation of indicators of urination. Ultrasound of the prostate gland. | Day 90
  Ultrasound of the prostate gland.
Evaluation of indicators of urination. Urofluometry. | Day 90
  Urofluometry.
Evaluation of indicators of urination. General urine analysis. | Day 90
  General urine analysis.
Evaluation of the inter-relapse period. Identification of an exacerbation of a chronic process. | Month 3
  Percentage of patients with exacerbation of chronic prostatitis and signs of disease recurrence during the follow-up period.
Evaluation of the inter-relapse period. Identification of signs of a relapse of the disease. | Month 3
  Percentage of patients with exacerbation of chronic prostatitis and signs of disease recurrence during the follow-up period.
Evaluation of the inter-relapse period. Identification of an exacerbation of a chronic process. | Month 6
  Percentage of patients with exacerbation of chronic prostatitis and signs of disease recurrence during the follow-up period.
Evaluation of the inter-relapse period. Identification of signs of a relapse of the disease. | Month 6
  Percentage of patients with exacerbation of chronic prostatitis and signs of disease recurrence during the follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Leonid Apanansky, Master, Study Director — SPP Pharmaclon Ltd.